CLINICAL TRIAL: NCT06394947
Title: Fluid Challenge in Intensive Care: a Worldwide Global Inception Cohort Study: The FENICE II Study
Brief Title: Fluid Challenge in Intensive Care The FENICE II Study
Acronym: FENICE II
Status: Completed | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: FENICE II
Record Dates: First submitted 2024-03-15; First posted 2024-05-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Critical Illness; Septic Shock
Keywords: Fluid Therapy; Fluid Challenge; Fluid Bolus; Intensive Care; Hemodynamic Monitoring
MeSH Terms: conditions — Critical Illness; Shock, Septic | interventions — Water-Electrolyte Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fluid administration (any type) — The fluid challenge (FC) (bolus) is defined as the administration of any bolus of fluid (crystalloid or colloid) which is expected to affect pressure/flow/perfusion variables. The FC is expected to be completed within 30 min.
  Other Names: Fluid Infusion; Fluid Bolus; Fluid Balance

SUMMARY:
Fluids are considered the primary treatment for critically ill patients admitted to the intensive care unit (ICU), aiming to replace losses and or to enhance venous return, stroke volume, and consequently, cardiac output and tissue oxygen delivery. The modalities, volumes, and targets employed to titrate fluid therapy vary significantly in current clinical practice, as shown by the original FENICE study 10 years ago. FENICE studied how fluid challenges are given at the bedside. Very little is known about how this practice has changed since, how fluid administration (maintenance) is performed in general, and how the modality may impact outcomes. FENICE II is designed to explore these issues.

Objectives:

To provide a comprehensive global description of fluid administration modalities during the initial days of ICU admission and to explore any association between fluid administration characteristics and clinical outcomes.

To describe the fluid challenge administration modality and appraise the use of variables and functional hemodynamic tests to guide bolus infusion.

DETAILED DESCRIPTION:
Primary aim: The primary aim is to describe the modality of fluid administration during the first 5 days of ICU stay considering 1) the overall fluid balance; 2) the characteristics of the fluids given; 3) the modality of fluid administration.

Secondary aims:

* To explore any association between fluid administration characteristics and clinical outcomes (see further)
* To evaluate factors potentially associated with the respective proportion of the different modalities of fluid administration
* To characterize FC administration modality in a large cohort of ICU patients.

Statistical Analysis:

Data will be described as median and interquartile range (IQR) or number and percentage. Categorical variables were compared using Fisher's exact test and continuous variables using the nonparametric Wilcoxon test, Mann-Whitney test, or Kruskal-Wallis test.

Volume of fluid and fluid balance (primary outcome) will be reported as median [IQR] from day 1 to day 5. This volume, fluid balance and respective volume of bolus and continuous fluid administration will be reported as distinct alluvial plots reporting median of fluid at day 1 to 5 per quartile along with outcome.

In way to assess relationship between volume of fluid received, characteristics and outcome (secondary outcome), longitudinal cluster modelling will be used to identify clusters of patients with similar patterns of fluid administration profile. Longitudinal k-mean will be used to assess change in fluid received each day from day 1 to day 3. In way to avoid misinterpretation of findings due to time dependent competing events such death or ICU discharge, this analysis will be performed on patients alive and still in the ICU at day 3. A sensitivity analysis will be performed during first 5 days on the subgroup of patients alive and not discharged during first 5 ICU-days.

In way to assess impact of fluid administration modality/strategy on outcome (secondary endpoint), factors associated with in-hospital mortality, including identified cluster of fluid administration, will be assessed using mixed logistic regression where in-hospital mortality will be event of interest. Center effect will be included as a random effect against the intercept.

For secondary outcomes, and in particular for day-30 mortality, number of days alive without vasopressors, mechanical ventilation or renal replacement therapy, will be assessed using survival analysis.

All tests will be two-sided, and P-value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

• All consecutive adult (≥18 years old) patients admitted to ICU and expected to stay at least 48h.

Exclusion Criteria:

* Planned admission after surgery for overnight ICU stay.
* Refusal of consent
* Moribund patients (i.e. expected survival < 24h)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult (≥18 years old) patients admitted to the intensive care unit and expected to stay at least 48h.
Sampling Method: Non-Probability Sample
Enrollment: 4734 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Composite of various aspects of fluid therapy | FIve days from ICU admission
  Modality of fluid administration during ICU stay considering 1) the overall fluid balance; 2) the characteristics of the fluids given; 3) the modality of fluid administration

SECONDARY OUTCOMES:
ICU mortality | Up to 30 days from ICU admission
  Mortality during ICU stay
In-hospital Mortality | Up to 30 days from ICU admission
  Mortality during hospital stay after ICU discharge
Alive without any organ support | between inclusion and 30 days later
  Number of calendar days between inclusion and 28 days that the patient is alive and with no requirement of cardiovascular, respiratory and renal support.
Organ Dysfunction - Lung | between inclusion and 30 days later
  Time to cessation of mechanical ventilation during ICU stay [The number of calendar days between intubation / start of mechanical ventilation and extubation / liberation from mechanical ventilation] (maintained for at least 48 hours)].
Organ Dysfunction - Heart | between inclusion and 30 days later
  Time to cessation of vasopressor support during ICU stay (The number of hours between enrollment and complete stopping of vasopressor support (defined as its complete interruption for at least 24 consecutive hours).
Organ Dysfunction - Renal | between inclusion and 5 days later
  Variation of creatinine-based KDIGO stage. Renal function assessed according to KDIGO staging system.
Organ Dysfunction - Renal | between inclusion and 30 days later
  Time to cessation of Renal Replacement during ICU stay [The number of calendar days between start of renal replacement therapy and complete liberation from renal replacement therapy (at least 48 hours for continuous replacement modalities and 5 days for intermittent ones).
Organ Dysfunction | between inclusion and 5 days later
  Variation of daily SOFA score.

OTHER OUTCOMES:
All aforementioned outcomes | 30 days from ICU admission
  Pre-defined subgroup analysis in patients admitted with septic shock
All aforementioned outcomes | 30 days from ICU admission
  Pre-defined subgroup analysis in patients admitted with neutropenia

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Humanitas Clinical and Research center, Rozzano, Milan
  - Humanitas Research Hospital, Milan

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Cecconi M, Hofer C, Teboul JL, Pettila V, Wilkman E, Molnar Z, Della Rocca G, Aldecoa C, Artigas A, Jog S, Sander M, Spies C, Lefrant JY, De Backer D; FENICE Investigators; ESICM Trial Group. Fluid challenges in intensive care: the FENICE study: A global inception cohort study. Intensive Care Med. 2015 Sep;41(9):1529-37. doi: 10.1007/s00134-015-3850-x. Epub 2015 Jul 11. PMID 26162676
- See also: Related Info — https://www.esicm.org/trials-group-2/fenice/